CLINICAL TRIAL: NCT01297933
Title: Intravenous Omega-3 Fatty Acid (Omegaven) for Pediatric Patients With Total Parenteral Nutrition Associated Liver Dysfunction
Brief Title: Compassionate Use of Omegaven for Pediatric Patients With Parenteral Nutrition Associated Liver Disease
Acronym: Omegaven
Status: Approved for marketing | Type: Expanded Access
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Maria Mascarenhas, Section Chief, Clinical Nutrition, Children's Hospital of Philadelphia
Other Study IDs: 10-007681
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Cholestasis; Short Bowel Syndrome
Keywords: parenteral nutrition associated liver disease; cholestasis; short bowel syndrome; Omegaven
MeSH Terms: conditions — Cholestasis; Short Bowel Syndrome | interventions — fish oil triglycerides

INTERVENTIONS:
Drug: Omegaven — 10% Omegaven 1g/kg/day, Intravenous by continuous infusion in conjunction with parenteral nutrition, until the patient no longer requires parenteral nutrition or until participation in the study is terminated.

SUMMARY:
A compassionate use protocol to provide Omegaven to pediatric patients with parenteral nutrition (PN) dependence and parenteral nutrition associated liver disease (PNALD).

DETAILED DESCRIPTION:
Omegaven is an intravenous fat emulsion (IFE) comprised of omega-3 fatty acids derived from fish oil. It will be used in an open label compassionate use treatment protocol, as an alternative to soybean oil (omega-6), as the sole IFE source of parenteral nutrition in an effort to reduce and/or reverse parenteral nutrition associated liver disease. The study will evaluate the safety and efficacy of Omegaven use in pediatric patients with PN dependence and PNALD.

ELIGIBILITY:
Inclusion Criteria:

* PN dependence due to congenital or acquired gastrointestinal disease
* Predicted PN requirement for at least an additional 30 days
* Parenteral nutrition associated liver disease (PNALD), defined as two conjugated bilirubin levels >= 2 mg/dL at least one week apart, must be obtained to demonstrate persistence of PNALD
* Failure to respond to standard therapies which may include cycling PN, reduction in the dose of soybean derived IFE, attempts to advance enteral feeds, ursodiol, metronidazole, and avoidance of excessive caloric provision
* signed parent or legal guardian informed consent

Exclusion Criteria:

* Acute treatable infection (e.g. urinary tract infection, sepsis)
* Known allergy to egg or fish protein
* Contraindications to Omegaven
* Pregnancy
* Serum triglyceride level greater than 400 mg/dL at baseline
* History of severe hemolytic disorders or INR greater than 1.5 at baseline (INR cutoff of greater than 2 for infants less than 1 week of age)

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Maria Mascarenhas, MBBS, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Alwayn IP, Gura K, Nose V, Zausche B, Javid P, Garza J, Verbesey J, Voss S, Ollero M, Andersson C, Bistrian B, Folkman J, Puder M. Omega-3 fatty acid supplementation prevents hepatic steatosis in a murine model of nonalcoholic fatty liver disease. Pediatr Res. 2005 Mar;57(3):445-52. doi: 10.1203/01.PDR.0000153672.43030.75. Epub 2005 Jan 19. PMID 15659701
- [Background] Diamond IR, Sterescu A, Pencharz PB, Kim JH, Wales PW. Changing the paradigm: omegaven for the treatment of liver failure in pediatric short bowel syndrome. J Pediatr Gastroenterol Nutr. 2009 Feb;48(2):209-15. doi: 10.1097/MPG.0b013e318182c8f6. PMID 19179884
- [Background] Gura KM, Parsons SK, Bechard LJ, Henderson T, Dorsey M, Phipatanakul W, Duggan C, Puder M, Lenders C. Use of a fish oil-based lipid emulsion to treat essential fatty acid deficiency in a soy allergic patient receiving parenteral nutrition. Clin Nutr. 2005 Oct;24(5):839-47. doi: 10.1016/j.clnu.2005.05.020. PMID 16029913
- [Background] Gura KM, Lee S, Valim C, Zhou J, Kim S, Modi BP, Arsenault DA, Strijbosch RA, Lopes S, Duggan C, Puder M. Safety and efficacy of a fish-oil-based fat emulsion in the treatment of parenteral nutrition-associated liver disease. Pediatrics. 2008 Mar;121(3):e678-86. doi: 10.1542/peds.2007-2248. PMID 18310188
- [Background] Puder M, Valim C, Meisel JA, Le HD, de Meijer VE, Robinson EM, Zhou J, Duggan C, Gura KM. Parenteral fish oil improves outcomes in patients with parenteral nutrition-associated liver injury. Ann Surg. 2009 Sep;250(3):395-402. doi: 10.1097/SLA.0b013e3181b36657. PMID 19661785
- [Background] Van Aerde JE, Duerksen DR, Gramlich L, Meddings JB, Chan G, Thomson AB, Clandinin MT. Intravenous fish oil emulsion attenuates total parenteral nutrition-induced cholestasis in newborn piglets. Pediatr Res. 1999 Feb;45(2):202-8. doi: 10.1203/00006450-199902000-00008. PMID 10022591